CLINICAL TRIAL: NCT01082718
Title: Pharmacokinetics of Mefloquine-Artesunate in Pregnant Women With Uncomplicated Plasmodium Falciparum Infection
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Logistical difficulties
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAACT PK
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Malaria; Pregnancy
Keywords: Malaria; Pregnancy; Pharmacokinetics; Brazil
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnant women (Experimental): Pregnant women with P. falciparum malaria
  Interventions: Drug: Mefloquine Artesunate
- Non pregnant women (Active Comparator): Non pregnant women with P. falciparum malaria
  Interventions: Drug: Mefloquine Artesunate

INTERVENTIONS:
Drug: Mefloquine Artesunate — Mefloquine-artesunate fixed dose combination (Farmanguinhos): Artesuanto 100 mg and Mefloquine 220mg per tablet, dosed once daily for 3 days such that mefloquine dose is approximately 8mg/kg/day.
  Other Names: Artesunato- mefloquina

SUMMARY:
Artemisinin-based combination therapies (ACTs) are now the treatment of choice for malaria in non-pregnant individuals living in areas with established chloroquine resistance; they have been shown to be both safe and highly efficacious. There is rapidly increasing experience with artemisinin derivatives in the 2nd and 3rd trimesters of pregnancy, with over 1,000 well documented cases with no reported serious adverse effects to mother or fetus (WHO Malaria Treatment Guidelines, 2006). Many countries in Latin America have abandoned the previous 1st line regimen of Quinine-Clindamycin for treatment of malaria in pregnancy, a complex and poorly tolerated regimen with low adherence, in favor of ACTs, despite limited safety and pharmacokinetic data on the use of these compounds in pregnant women. Lack of pharmacokinetic data may lead to underdosing of pregnant women, with subsequent reduced efficacy and increased potential for development of resistance.

One ACT regimen, Artesunate-Mefloquine, has been developed as a fixed-dose combination (Farmanguinhos Artesunato + Mefloquina), as part of an international collaborative research effort led by Drugs for Neglected Diseases Initiative (DNDi), and manufactured by Farmanguinhos, laboratory of the Brazilian Ministry of Health. Initial clinical trials suggest that it is very well tolerated and efficacious in both pregnant and non-pregnant individuals. The convenient dosing afforded by a fixed drug combination make this a very promising candidate for treatment of pregnant women with malaria. Preliminary pharmacokinetic data from mefloquine monotherapy and prophylaxis suggest that the peak concentration of mefloquine is lowered in pregnant women. Prior to wide-spread adoption of the Artesunate-Mefloquine combination, further studies on safety, efficacy, and dose optimization are imperative. We propose to compare the pharmacokinetics of the fixed combination of mefloquine-artesunate (MA) for treatment of P.falciparum in 28 pregnant women in the second and third trimesters to the pharmacokinetics of this regimen in 28 matched non-pregnant P.falciparum infected women. This will allow us to determine whether the standard adult dose is sufficient for pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Cases: Pregnant women, age ≥18 years, in 2nd or 3rd trimester (gestational age ≥12 weeks determined by LMP and confirmed by fundal height measurement) Controls: Non-pregnant women ≥18 years old (negative urine pregnancy test)
2. Presence of P. falciparum ≤ 50,000 parasites/microliter
3. Fever (≥37.5C) or history of fever in preceding 48 hours
4. Willing to sign or thumb print informed consent
5. Willing to be hospitalized for 3 days and to return for scheduled follow up visits for treatment and observation until delivery
6. Willing to deliver in health facility

Exclusion Criteria:

1. Pregnancy < 12 weeks
2. Presence of malaria species other than P. falciparum on the slide (P. vivax, P. malariae, or P. ovale, or mixed infection (P. falciparum in combination with any other malaria species)
3. History of allergy or hypersensitivity to interventional drugs
4. Exposure to antimalarial drugs and other drugs with antimalarial activity within the past 2 months, as determined by history from the woman.
5. Patients taking drugs with possible interaction with study drugs (ie, digoxin or warfarin)
6. History or family history of epilepsy or psychiatric disorder
7. Presence of signs and symptoms of severe malaria
8. Inability to tolerate oral medication (repeated vomiting, impairment of consciousness). Vomiting of any of the treatment doses will lead to exclusion from the pharmacokinetic sampling, but not the follow-up for drug efficacy.
9. History of chronic disease including diabetes, renal failure, hepatic failure, heart disease requiring anti-arrhythmic drugs or warfarin, AIDS (HIV itself will not be an exclusion, but anyone with AIDS or HIV requiring HAART will be excluded), hemoglobinopathy,
10. Participant's inability to return for follow up visits
11. Age <18 years
12. Hb<8g/dl

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of Mefloquine - artesunate in pregnant versus matched non-pregnant women with P. falciparum malaria | Multiple measures up to 63 days

SECONDARY OUTCOMES:
PCR correct cure rate on Day 63 | Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Meghna Desai, MPH PhD, Principal Investigator — Centers for Disease Control and Prevention